CLINICAL TRIAL: NCT01927666
Title: A Human Intervention Trial Investigating the Conversion of Encapsulated Glucoraphanin to Isothiocyanates; and the Potential Link Between the Extent of the Conversion to an Individual's Gut Microbiota Phylogeny and Genotype.
Brief Title: The Conversion of ENcapsulated GlucorAphanin, Gut Microbiota Phylogeny and gEnotype Study (ENGAGE)
Acronym: ENGAGE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Quadram Institute Bioscience (Other)
Collaborators: Biotechnology and Biological Sciences Research Council (Other); The Danish Council for Strategic Research (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 12/EE/0483
Record Dates: First submitted 2013-08-20; First posted 2013-08-22 (Estimated); Last update posted 2016-09-05 (Estimated); Status verified 2015-11

CONDITIONS: Healthy
Keywords: glucoraphanin; broccoli; gut microbiota
MeSH Terms: interventions — glucoraphanin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- dietary intervention (Experimental): To measure the variation in extent of ITC excretion in urine from a capsule delivered dose of 100mg glucoraphanin
  Interventions: Dietary Supplement: 100mg glucoraphanin

INTERVENTIONS:
Dietary Supplement: 100mg glucoraphanin — The extent of ITC excretion in urine from a capsule delivered dose of glucoraphanin

SUMMARY:
The variation in extent of isothiocyanate (ITC) excretion in urine from a capsule delivered dose of glucoraphanin will correlate with differences in (a) the gut microbiota, and (b) the genotype of key polymorphic genes (GSTM1, GSTT1, and other as yet undetermined candidate genes).

Our study is a human dietary intervention in which participants will consume one capsule containing 100mg purified glucoraphanin from broccoli. The levels of glucoraphanin delivered by the capsule are similar to one to two portions of broccoli. As this is purified glucoraphanin there is no myrosinase enzyme present. All conversion of the glucoraphanin, contained within the capsule, to ITC will therefore occur by enzymes found in the gut microbiota.

The ability of the glucoraphanin in the capsule to be metabolised to ITCs by the gut microflora is unknown and will be assessed by measuring ITCs excreted in the urine. The ITCs will be quantified in urine using validated analytical methods.

It has been shown in human dietary intervention studies that the extent of conversion of glucosinolates varies greatly. In order to assess possible causative factors for variation in rate of glucoraphanin metabolism each participant will provide a faecal sample from which their faecal gut microbiota phylogeny will be analysed.

For a small number of participants a second faecal sample will be requested (a maximum of 3 participants). It is our aim to select one low, one medium and one high ITC excreter. Ideally the low and high excreters would be within the lowest and highest 5% excretion of ITC and the third participant would be as close to the mean ITC excretion as possible. The aim would be to culture the faecal microbiota over time with repeat dosing of glucoraphanin in order to select for microbiota that are able to metabolise glucoraphanin. It is known that the main hydrolysis product of glucoraphanin, sulforaphane, has a variety of benefits to human health, however there is no known clinical relevance to being a high, medium or low excreter of ITC.

For each participant a blood sample will also be requested in order that we can assess whether genotype affects the rate of ITC excretion in urine. The GSTM1 genotype and other, as yet, unidentified candidate genes of each participant will be determined. Whether the genotype affects the rate of ITC excretion either alone or in combination with the phylogenetic profile will be assessed.

DETAILED DESCRIPTION:
Glucosinolates (GSLs) are non-volatile sulphur-containing phytochemicals (secondary metabolites) found in plant tissues of cruciferous crops, such as broccoli, cabbage and watercress. Glucosinolates accumulate in these foods with glucoraphanin being the predominant glucosinolate found in broccoli. When tissue is disrupted the glucosinolates are converted to isothiocyanates (ITCs) by the enzyme myrosinase. Sulforaphane is the predominant ITC obtained by enzymatic hydrolysis from glucoraphanin. When vegetables are cooked very thoroughly the myrosinase enzyme is denatured which results in GSLs passing through the gastrointestinal (GI) tract into the colon.

The ITCs have been shown in animal studies to exert diverse biological effects, such as anti-oxidant effects; anti-inflammatory properties; inhibition of platelet aggregation; reduction of systolic blood pressure and the reduction of cholesterol levels; all of which reduce the risk developing cardiovascular diseases. Sulforaphane has been linked to health benefits in humans, such as cancer chemoprevention and helping to maintain a healthy heart.

When cooked cruciferous vegetables, in which the myrosinase enzyme has been inactivated, are consumed, some of the microflora in the colon produce a myrosinase-like enzyme that can also convert glucosinolates to ITCs. This process of gut microbiota conversion of glucoraphanin to ITC is abolished by enteric antibiotics and bowel cleansing. There have been several in vitro studies performed with both pure and mixed cultures of bacteria confirming the ability of bacterial strains found within the human gut having the ability to metabolize GSLs in culture. It has been shown that the extent of conversion of GSLs to ITCs by human gut microbiota varies greatly between individuals but the conversion rate from repeated determinations within individuals are much more consistent. A recent study attempted to correlate the conversion of glucosinolate ex vivo by human gut bacteria to in vivo data of glucosinolate metabolism from a small number of individuals, however no specific link to individual bacterial specials was established.

Our study is a human dietary intervention in which participants will consume one capsule containing 100mg purified glucoraphanin from broccoli. The levels of glucoraphanin delivered by the capsule are similar to one to two portions of broccoli. As this is purified glucoraphanin there is no myrosinase enzyme present. All conversion of the glucoraphanin, contained within the capsule, to ITC will therefore occur by enzymes found in the gut microbiota.

The ability of the glucoraphanin in the capsule to be metabolised to ITCs by the gut microflora is unknown and will be assessed by measuring ITCs excreted in the urine. In brief each participant on the study will be requested to abstain from any glucosinolate and ITC containing foods for three days prior to dietary intervention, and for a further 24 hours during the intervention. They will be requested to fast overnight prior to the study day intervention and on the morning after the fast collect a urine sample. This will effectively constitute a negative control sample and be used as a measure of compliance with the dietary restriction. The participant will then be given the glucoraphanin capsule along with their breakfast. The dietary restriction will continue for a further 24hours, during which time the participant will collect all the urine they produce. The ITCs will be quantified in urine by HP-LC and LC-MS using validated analytical methods. Once the 24 hour urine collection is complete the dietary restriction will cease.

It has been shown in human dietary intervention studies that the extent of conversion of glucosinolates varies greatly. In order to assess possible causative factors for variation in rate of glucoraphanin metabolism each participant will provide a faecal sample from which their faecal gut microbiota phylogeny will be analysed. A detailed description of how the sample should be collected along with all equipment necessary will be provided. The faecal samples will be returned to the study scientist within two hours of production in order to maintain faecal bacteria viability.

For a small number of participants a second faecal sample will be requested (a maximum of 3 participants). The aim is to select one low, one medium and one high ITC excreter. Ideally the low and high excreters would be within the lowest and highest 5% excretion of ITC and the third participant will be as close to the mean ITC excretion as possible. The aim is to culture the faecal microbiota over time with repeat dosing of glucoraphanin in order to select for microbiota that are able to metabolise glucoraphanin. It is known that the main hydrolysis product of glucoraphanin, sulforaphane, has a variety of benefits to human health, however there is no known clinical relevance to being a high, medium or low excreter of ITC.

Several epidemiological and intervention studies suggest that the health benefits and physiological response to cruciferous vegetables may be mediated by an individual's GSTM1 genotype (glutathione-S-transferases (GST) gene family). When ITCs are absorbed into the body, they conjugate with glutathione and are then metabolised through the mercapturic acid pathway. Conjugation happens spontaneously due to the relatively high concentration of glutathione within cells compared to the ITC concentration. However as non-conjugated ITCs occur in the plasma, at some stage there must be dissociation of the ITC-thiol conjugate. It is thought that this may be catalyzed by the GSTM1 enzyme. Approximately 50% of the population have a homologous deletion of the GSTM1 gene resulting in a null genotype, and 20% has a deletion of the GSTT1 gene. There are some studies, including one of our own, that suggests that GSTM1 genotype may affect the rate of ITC excretion in urine, but have not suggested that GSTM1 genotype affects the peak plasma ITC concentration.

Unpublished results from a previous intervention, the Diet and Vascular Health study; Clinical Trials.gov: NCT01114399 have added credence to the notion that GSTM1 nulls metabolise sulforaphane in a different manner to those with a functional GSTM1 allele. Along with the GST gene family and their association with cruciferous vegetables there may be other genes of interest that may be able to determine the extent of glucoraphanin conversion to sulforaphane. Work carried out on our previous intervention, the Diet and Vascular Health study has sought to investigate possible candidate genes. With a substantial amendment looking to take a more global approach in identifying candidate genes of interest by performing an Affymetrix SNP analysis on samples from participants who had been on a high glucoraphanin diet.

Therefore the GSTM1 genotype and other, as yet, unidentified candidate genes of each participant will be determined to assess whether genotype affects the rate of ITC excretion in urine, either alone, or in combination with their phylogenic profile. A 5 ml blood sample will be taken from each participant and the DNA extracted, PCR will then be used to test whether the gene is present or not.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged 18 or over
* Smokers and non-smokers
* Those that live within 40 miles, and 2 hours travelling time, of Norwich

Exclusion Criteria:

* Women who are or have been pregnant within the last 12 months or breast feeding.
* Those currently suffering from or have ever suffered from any gastrointestinal disease, gastrointestinal disorders and/or surgery including regular diarrhoea and constipation (excluding hiatus hernia unless symptomatic) or study intervention/procedure is contraindicated.
* Have been diagnosed with any long-term medical condition that may affect the study outcome (e.g. diabetes, haemophilia, cardiovascular disease, glaucoma, anaemia). These will be assessed on an individual basis.
* On medication that may affect the study outcome.
* Those that have used antibiotics within the previous one month or on long-term antibiotic therapy.
* Those regularly taking laxatives (once a month or more)
* Those intermittently using pre &/or pro biotics unless willing to abstain for 1 month prior and during study period. (If used regularly (3+ times a week, and for more than one month) and will continue throughout study period then do not exclude).
* Those taking dietary supplements or herbal remedies which may affect the study outcome -unless the participant is willing to discontinue taking them for 1 month prior to starting study. Please note that some supplements may not affect the study and this will be assessed on an individual basis
* Regular/ recent (within 3 months) use of colonic irrigation or other bowel cleansing techniques.
* Parallel participation in another research project which involves dietary intervention and/or sampling of blood
* Any person related to or living with any member of the study team
* Participation in another research project which involves blood sampling within the last four months unless total blood from both studies does not exceed 470mL
* are unwilling to provide GPs contact details
* are unable to provide written informed consent
* are not suitable to take part in this study because of your screening results
* have donated or intend to donate blood within 16 weeks of the first and last study samples
* Those with a body mass index (BMI, kg/m2) <20
* Those who are unable to swallow capsules
* Those who do not have access to a freezer

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2012-12; Primary Completion 2014-12 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Urinary ITC concentration | In 24h collections at (i) baseline and (ii) following glucoraphanin capsule administration.
  To measure urinary ITC by HP-LC and LC-MS using validated methods in urine collected during a dietary restriction period both before and after (24 hour urine collection) consumption of a 100mg glucoraphanin capsule.

SECONDARY OUTCOMES:
Faecal microbiota phylogenetic analysis | At baseline
  To measure gut microbiota populations by faecal bacteria phylogenetic analysis.
Genotype | At baseline
  To determine the genotype of participants for key polymorphic genes by PCR on DNA extracted from blood.

CONTACTS AND LOCATIONS:
Overall Officials: Richard Mithen, PhD, Principal Investigator — Quadram Institute Bioscience
Locations (1):
- Institute Of Food Research, Norwich, Norfolk, United Kingdom

REFERENCES:
- [Background] Armah CN, Traka MH, Dainty JR, Defernez M, Janssens A, Leung W, Doleman JF, Potter JF, Mithen RF. A diet rich in high-glucoraphanin broccoli interacts with genotype to reduce discordance in plasma metabolite profiles by modulating mitochondrial function. Am J Clin Nutr. 2013 Sep;98(3):712-22. doi: 10.3945/ajcn.113.065235. PMID 23964055